CLINICAL TRIAL: NCT03922815
Title: Influence of Adequacy of Anaesthesia Monitoring on Both Operators' and Patients' Satisfaction in Patients Undergoing Colonoscopic Procedures
Brief Title: Adequacy of Anaesthesia for Colonoscopic Procedures
Acronym: AoAColon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SilesianMUKOAiIT12
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2018-10

CONDITIONS: Colonic Diseases, Functional
Keywords: Surgical Pleth Index (SPI); Adequacy of Anaesthesia (AoA); State Entropy (SE); Postoperative nausea and vomitting (PONV); Colonoscopy
MeSH Terms: conditions — Colonic Diseases, Functional; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Neither participant nor colonoscopic procedure provider are aware of the type of monitoring utilised during procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- haemodynamic parametres-guided deep sedation (Experimental): propofol will be tirtrated in a single dose of 0,5 mg/kg of body weight to disappearance of cilliary reflex; in the case of heart rate and/or arterial blood pressure increase by 20% a rescue dose of fentanyl 0,5 mcg per kilogram of body weight will be administered
  Interventions: Drug: rescue fentanyl; Drug: rescue propofol
- SE-guided propofol-fentanyl deep sedation (Experimental): propofol will be tirtrated in a single dose of 0,5 mg/kg of body weight to a target SE < 80 alongside with a rescue dose 0,5 mcg per kilogram of body weight of fentanyl in the case of heart rate and/or arterial blood pressure increase by 20%
  Interventions: Drug: rescue fentanyl; Drug: rescue propofol
- AoA-guided propofol-fentanyl deep sedation (Experimental): propofol will be tirtrated in a single dose of 0,5 mg/kg of body weight to a target SE < 80 alongside with a rescue dose 0,5 mcg per kilogram of body weightof fentanyl in the case of increase of SPI value > delta 15
  Interventions: Drug: rescue fentanyl; Drug: rescue propofol

INTERVENTIONS:
Drug: rescue fentanyl — a rescue dose of fentanyl 0,5 mcg per kilogram of body
  Other Names: rescue analgesia
Drug: rescue propofol — propofol in a single dose of 0,5 mg/kg of body weight
  Other Names: rescue sedation

SUMMARY:
The aim of this randomized prospective trial is to assess the utility of Adequacy of Anaesthesia technique (Response Entropy and Surgical Pleth Index) for monitoring pain perception intraoperatively and its influence on postoperative pain perception, both patients' and operators' satisfaction in patients undergoing colonoscopic procedures under intravenous sedation using propofol and fentanyl.

DETAILED DESCRIPTION:
Surgical Pleth Index (SPI) is reported to properly reflect nociception-antinociception balance in patients undergoing surgical procedures, where a value of 100 corresponds to a high stress level and a value of 0 to a low stress level; values near 50 or increase in value > delta 10 correspond to the stress level which is known to reflect requirement for rescue analgesia.

The applicability of SPI- guided deep sedation regimen in colonoscopic procedures has not been previously studied. Additionally, depth of sedation markedly influences the nociception-antinociception balance so its monitoring also proved useful in procedures performed under deep sedation.

Therefore, we aim to investigate if both SPI-guided fentanyl administration alongside with State Entropy guided propofol aministration (Adequacy of Anaesthesia monitoring) versus State Entropy guided propofol aministration alongside with fentanyl titration based on haemodynamic parametres versus fentanyl titration based on haemodynamic parametres only influence both patients' or operator's satisfaction from anaesthetic management.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo deep sedation for colonoscopic procedure
* general heath condition I-III of American Society of Anaesthesiology

Exclusion Criteria:

* necessity of administration of vasoactive drugs influencing SPI monitoring
* pregnancy
* anatomical malformation that make monitoring using SE sensor impossible
* general atherosclerosis, heart rhythm disturbances impairing SPI monitoring
* chronic medication using opioid drugs leading to resistancy to opioids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
intraoperative pain perception: 11 points numeric rating scale | after 2 hours after emergence from sedation
  the patient will be asked if he/she had any reminiscence of pain perception during procedure of colonoscopy using 11 points numeric rating scale (0 - no pain, 10 - maximum pain)
postoperative pain perception: 11 points numeric rating scale | immediately after emergence form sedation
  the patient will be asked if he/she had any pain perception after emergence from sedation after procedure of colonoscopy using 11 points numeric rating scale (0 - no pain, 10 - maximum pain)

SECONDARY OUTCOMES:
patient's satisfaction: 4 points numeric rating scale | 2 hours after emergence from sedation
  the patient will be asked if he/she was satisfied with sedation quality for the procedure of colonoscopy using 4 points numeric scale
operator's satisfaction: 4 points numeric scale | immediately after the end of the procedure
  the operator will be asked if he/she was satisfied with sedation quality for the procedure of colonoscopy using 4 points numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Michał J Stasiowski, M.D, Principal Investigator — Medical University of Silesia
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
article in AiIT 2019
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: on a reasonable request

REFERENCES:
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Result] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Result] Won YJ, Lim BG, Lee SH, Park S, Kim H, Lee IO, Kong MH. Comparison of relative oxycodone consumption in surgical pleth index-guided analgesia versus conventional analgesia during sevoflurane anesthesia: A randomized controlled trial. Medicine (Baltimore). 2016 Aug;95(35):e4743. doi: 10.1097/MD.0000000000004743. PMID 27583920
- [Result] Abu Baker F, Mari A, Aamarney K, Hakeem AR, Ovadia B, Kopelman Y. Propofol sedation in colonoscopy: from satisfied patients to improved quality indicators. Clin Exp Gastroenterol. 2019 Feb 26;12:105-110. doi: 10.2147/CEG.S186393. eCollection 2019. PMID 30881077
- [Result] Zhang W, Zhu Z, Zheng Y. Effect and safety of propofol for sedation during colonoscopy: A meta-analysis. J Clin Anesth. 2018 Dec;51:10-18. doi: 10.1016/j.jclinane.2018.07.005. Epub 2018 Jul 27. PMID 30059837